CLINICAL TRIAL: NCT06150417
Title: Metastasis-directed Radiotherapy (MDRT) for Men With De-novo Oligometastatic Prostate Cancer Treated With Long-term Androgen Deprivation Therapy in the STAMPEDE Trial (METANOVA)
Brief Title: MDRT in Prostate Cancer Treated With Long-term Androgen Deprivation Therapy in the STAMPEDE Trial (METANOVA)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE5823; U01CA257638 (NIH)
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer; Malignant Neoplasm of Prostate; Secondary Malignant Neoplasm of Prostate
Keywords: Metastasis-directed Radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists; Radiotherapy

STUDY DESIGN:
Intervention Model Description: Phase II non-blinded randomized study evaluating men with de novo oligometastatic prostate cancer randomized (1:1) to standard of care (SOC) versus SOC plus MDRT.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (Active Comparator): * Participants will receive the standard of care. Standard systemic therapy (SST) and definitive local therapy (radiotherapy [RT] or radical prostatectomy [RP]) are the standard of care for de novo oligometastatic prostate cancer. This arm will be used to compare to the experimental arm.
  * SST will begin 6 weeks of randomization and occur for 12 months. The definitive local therapy will be RT, with a small portion undergoing RP. Local therapy should be completed by the end of Week 20.
  Interventions: Drug: Androgen deprivation therapy (ADT); Drug: Androgen receptor signaling inhibitor (ARSI); Other: Local Therapy: Radical Prostatectomy (RP) or Radiotherapy (RT)
- SOC + MDRT (Experimental): * Participants will receive the standard of care. Standard systemic therapy (SST) and definitive local therapy (radiotherapy [RT] or radical prostatectomy [RP]) are the standard of care for de novo oligometastatic prostate cancer. This arm will be used to compare to the experimental arm.
  * SST will begin 6 weeks of randomization and occur for 12 months. The definitive local therapy will be RT, with a small portion undergoing RP. Local therapy should be completed by the end of Week 20.
  * MDRT should be completed by the end of Week 24. Depending on the participant, there are different approaches to MDRT dosing and fraction size.
  Interventions: Drug: Androgen deprivation therapy (ADT); Drug: Androgen receptor signaling inhibitor (ARSI); Other: Local Therapy: Radical Prostatectomy (RP) or Radiotherapy (RT); Radiation: Metastasis directed radiotherapy (MDRT)

INTERVENTIONS:
Drug: Androgen deprivation therapy (ADT) — Standard androgen deprivation therapy (ADT) will be administered at the discretion of treating physician.
Drug: Androgen receptor signaling inhibitor (ARSI) — Standard androgen receptor signaling inhibitors (ARSI) will be administered at the discretion of the treating physician.
Other: Local Therapy: Radical Prostatectomy (RP) or Radiotherapy (RT) — Local therapy will either be radiotherapy (RT) or radical prostatectomy (RP).
  * Prostate +/- pelvic nodal radiation
  * Radical prostatectomy + pelvic lymph node dissection
Radiation: Metastasis directed radiotherapy (MDRT) — In participants randomized to the MDRT arm, MDRT to all lesions will be performed by the end of Week 24. Selection of a particular regimen (the dose and fractionation) will based on the size and location of the participant's metastatic site and the surrounding normal tissue constraints.
  Arms: SOC + MDRT

SUMMARY:
The purpose of this study is to find out if giving radiation therapy (RT) to areas of metastatic prostate cancer at the time a participant is diagnosed will help control disease better than the usual treatment. This treatment is called metastasis-directed radiotherapy (MDRT).

The usual treatment for prostate cancer that has spread to other parts of the body is to give lifelong treatment with hormone therapy (also known as androgen deprivation therapy or ADT). Participants may also be given prostate RT even if the disease is metastatic. Participants will receive hormone therapy (the standard treatment for prostate cancer) for 12 months. The hormone therapy agents may be taken by mouth or given as an injection. Participants will also have prostate RT. Up to 50 participants will have surgery to remove the prostate instead of having prostate RT. A portion of the participants will be randomized to receive MDRT to areas where the cancer has spread. For participants who have surgery to remove their prostate, they will be asked to allow tissue samples collected during the surgery to be sent to an outside lab for research tests and extra blood samples drawn for research tests before starting the study, and at the time the cancer becomes worse if applicable. Participation in the study will last approximately 12 months, and will be followed by their doctor for up to five years per standard of care.

The main goal is to compare the efficacy of the standard of care (standard systemic therapy + definitive prostate-directed local therapy) versus the standard of care with metastasis-directed radiotherapy (MDRT) for consolidation of metastatic disease.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is the most common cancer in men worldwide, with 10% diagnosed with metastatic disease at the time of presentation. The metastatic capacity of cancers behaves along a spectrum of disease progression, such that some solid tumors have spread widely before clinical detectability and others never metastasize. While metastatic disease has historically been treated with palliative intent, an oligometastatic state where metastases are limited in number and location has emerged in which participants with oligometastatic disease may benefit from effective local therapy in addition to systemic therapy. Systemic standard-of-care therapies often include androgen deprivation therapy (ADT) and Androgen receptor signaling inhibitor (ARSI). Studies have shown that administering local radiotherapy (RT) to the prostate in addition to standard of care may improve radiographic profession-free survival. It may be even more efficacious to add metastasis-directed radiotherapy (MDRT) to the treatment of oligometastatic prostate cancer cases. More research is necessary to investigate the application of MDRT to improve disease control.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 years of age.
* Participant must have an ECOG performance status ≤ 1.
* Histologic confirmation of prostate adenocarcinoma of the prostate gland, with evidence of metastasis on imaging by conventional imaging (MRI, CT, or 99mTc bone scan) or PSMA PET/CT. Biopsy of sites of metastasis is strongly encouraged, but not required.

  * There must be at least 10-15 unstained slides from 2 cores of the highest tumor cellularity available.
* Newly diagnosed disease with no prior treatment(surgery, radiation or systemic treatment, ie hormone therapy or chemotherapy) to the primary disease.

  * Participants may have started LHRH agonist or antagonist therapy, and/or androgen receptor signaling inhibitor (ARSI) as long as it was not started more than 30 days before the participant is enrolled on this study.
* In participants who undergo only conventional imaging, oligometastatic disease is defined as 1-5 discrete metastatic sites in the bone and/or extra-pelvic lymph node (LN) stations.

  * Extra-pelvic LN stations are superior to the regional/pelvic LN stations. Pelvic LN stations commence at the bifurcation of the aorta and bifurcation of the proximal inferior vena cava to the common iliac veins.

    * Radiographic criteria for a LN to be considered a metastatic focus is defined as short-axis diameter in the axial plane of ≥ 1.0 cm, with irregular border and/or heterogeneous morphology
* In participants who undergo PSMA PET/CT (in the presence or absence of conventional imaging), oligometastatic disease is defined as 1-10 PSMA avid bone lesions and/or extra-pelvic LN stations. The MI-RADS reporting system will be followed to guide PSMA PET interpretation

  * In participants extra-pelvic nodal (M1a) disease only by PSMA PET/CT and M0 by conventional imaging (i.e. extra-pelvic LN did not meet size criteria by CT), participant must meet 2 of 3 following criteria in order to be eligible:

    * 1. PSA ≥ 40
    * 2. Evidence of cN1 disease (pelvic LN)
    * 3. Decipher score ≥ 0.89
* Adequate organ and marrow function to receive treatment per treating physician
* Medically fit for treatment and agreeable to follow-up.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

Participants with the presence of any of the following:

* Castration resistant prostate cancer (CRPC).
* Evidence of visceral or intracranial metastases.
* Participant receiving any other investigational agents for cancer.
* Participant is participating in a concurrent treatment protocol for cancer.
* Unable to lie flat during or tolerate PET/MRI, PET/CT or SBRT.
* Prior definitive treatment to the primary prostate cancer or pelvis.
* Participant with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled diabetes (HgA1c > 10), active pituitary or adrenal dysfunction, or psychiatric illness/social situations that would limit compliance with study requirements
* History of another active malignancy within the previous 2 years, except for non-melanoma skin cancer, non-muscle invasive bladder cancer, or a malignancy that is considered cured with minimal risk of recurrence
* Active Crohn's disease or ulcerative colitis despite medical management.
* Refusal to sign informed consent.
* Any condition that in the opinion of the investigator would preclude participation in this study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival (FFS) | Up to 5 years from treatment
  Failure-free survival, defined as time from randomization to first evidence of at least one of: biochemical failure; progression either locally in lymph nodes, or in distant metastases; skeletal related event (where confirmed disease progression);any salvage intervention (local or systemic) required after 12m of planned SOC therapy; or death from prostate cancer.
  Biochemical failure, based on the PSA nadir in the first 24 weeks after randomization, is defined as at least one of:
  post-RT:
  1. as per the Prostate Cancer Clinical Trials Working Group 3 (PCWG3), where PSA must rise by ≥ 25% and ≥ 2ng/mL above nadir, confirmed by progression at two time points at least 3 weeks apart
  2. post-RP: serum PSA nadir + 0.4 ng/mL, requiring confirmation ≥4 weeks later

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 5 years from treatment
  Overall Survival (OS) is defined as the time from randomization until death due to any cause. For participants who survive, time to death will be censored at the time of last contact. The distributions of OS for each treatment arm will be plotted using the Kaplan-Meier method, and median values for each will be estimated and reported with 95% CIs for each treatment arm and compared using stratified log-rank tests. Univariable Cox proportional hazard models will be used to estimate the effect of MDRT on OS.
Radiographic progression-free survival (rPFS) | Up to 5 years from treatment
  Radiographic progression-free survival (rPFS) is defined as the time from randomization until clinical progression, detection of at least one new metastatic lesion on CT, MRI, bone scan or Prostate Specific Membrane Antigen (PSMA) PET, or death from prostate cancer. The distributions of rPFS for each treatment arm will be plotted using the Kaplan-Meier method, and median values for each will be estimated and reported with 95% CIs for each treatment arm and compared using stratified log-rank tests. Univariable Cox proportional hazard models will be used to estimate the effect of MDRT on rPFS.
Time-to-next-intervention (TTNI) | Up to 5 years from treatment
  TTNI is defined as time-to-next-intervention. TTNI will be summarized in each arm and compared using Chi-square tests, as well as time-to-event analyses using cumulative incidence methods.
Time-to-castration-resistant prostate cancer | Up to 5 years from treatment
  The rate of time-to-castration-resistant prostate cancer will be summarized in each arm and compared using Chi-square tests, as well as time-to-event analyses using cumulative incidence methods.
Prostate-specific cancer mortality (PCSM) | Up to 5 years from treatment
  Prostate cancer specific mortality (PCSM) is defined the time from randomization to death directly attributable to prostate cancer, death from treatment complications, or death from unknown causes in participants with active prostate cancer or previously documented clinical or biochemical relapse.
Change in EPIC-26 Sexual Domain Score | Baseline, 1 year after treatment
  EPIC-26 is the validated short version of "The Expanded Prostate Cancer Index Composite". EPIC-26 will be administered as a health related quality of life questionnaire for participants with prostate cancer. EPIC-26 consists of 26 items under 5 domains. This study will analyze 4 of the domains, including the urinary, bowel, sexual, and hormonal domain. Each domain will be scaled, scored, and compared by arm.
  EPIC-26 assess participant function and bother on a qualitative scale which is then normalized on a scale of 0 to 100 (worst to best) to calculate individual domain scores.
Change in EPIC-26 Sexual Domain Score | Baseline, 3 years after treatment
  EPIC-26 is the validated short version of "The Expanded Prostate Cancer Index Composite". EPIC-26 will be administered as a health related quality of life questionnaire for participants with prostate cancer. EPIC-26 consists of 26 items under 5 domains. This study will analyze 4 of the domains, including the urinary, bowel, sexual, and hormonal domain. Each domain will be scaled, scored, and compared by arm.
  EPIC-26 assess participant function and bother on a qualitative scale which is then normalized on a scale of 0 to 100 (worst to best) to calculate individual domain scores.
Change in EPIC-26 Urinary Domain Score | Baseline, 1 year after treatment
  EPIC-26 is the validated short version of "The Expanded Prostate Cancer Index Composite". EPIC-26 will be administered as a health related quality of life questionnaire for participants with prostate cancer. EPIC-26 consists of 26 items under 5 domains. This study will analyze 4 of the domains, including the urinary, bowel, sexual, and hormonal domain. Each domain will be scaled, scored, and compared by arm.
  EPIC-26 assess participant function and bother on a qualitative scale which is then normalized on a scale of 0 to 100 (worst to best) to calculate individual domain scores.
Change in EPIC-26 Urinary Domain Score | Baseline, 3 years after treatment
  EPIC-26 is the validated short version of "The Expanded Prostate Cancer Index Composite". EPIC-26 will be administered as a health related quality of life questionnaire for participants with prostate cancer. EPIC-26 consists of 26 items under 5 domains. This study will analyze 4 of the domains, including the urinary, bowel, sexual, and hormonal domain. Each domain will be scaled, scored, and compared by arm.
  EPIC-26 assess participant function and bother on a qualitative scale which is then normalized on a scale of 0 to 100 (worst to best) to calculate individual domain scores.
Change in EPIC-26 Hormone Domain Score | Baseline, 1 year after treatment
  EPIC-26 is the validated short version of "The Expanded Prostate Cancer Index Composite". EPIC-26 will be administered as a health related quality of life questionnaire for participants with prostate cancer. EPIC-26 consists of 26 items under 5 domains. This study will analyze 4 of the domains, including the urinary, bowel, sexual, and hormonal domain. Each domain will be scaled, scored, and compared by arm.
  EPIC-26 assess participant function and bother on a qualitative scale which is then normalized on a scale of 0 to 100 (worst to best) to calculate individual domain scores.
Change in EPIC-26 Hormone Domain Score | Baseline, 3 years after treatment
  EPIC-26 is the validated short version of "The Expanded Prostate Cancer Index Composite". EPIC-26 will be administered as a health related quality of life questionnaire for participants with prostate cancer. EPIC-26 consists of 26 items under 5 domains. This study will analyze 4 of the domains, including the urinary, bowel, sexual, and hormonal domain. Each domain will be scaled, scored, and compared by arm.
  EPIC-26 assess participant function and bother on a qualitative scale which is then normalized on a scale of 0 to 100 (worst to best) to calculate individual domain scores.
Change in EPIC-26 Bowel Domain Score | Baseline, 1 year after treatment
  EPIC-26 is the validated short version of "The Expanded Prostate Cancer Index Composite". EPIC-26 will be administered as a health related quality of life questionnaire for participants with prostate cancer. EPIC-26 consists of 26 items under 5 domains. This study will analyze 4 of the domains, including the urinary, bowel, sexual, and hormonal domain. Each domain will be scaled, scored, and compared by arm.
  EPIC-26 assess participant function and bother on a qualitative scale which is then normalized on a scale of 0 to 100 (worst to best) to calculate individual domain scores.
Change in EPIC-26 Bowel Domain Score | Baseline, 3 years after treatment
  EPIC-26 is the validated short version of "The Expanded Prostate Cancer Index Composite". EPIC-26 will be administered as a health related quality of life questionnaire for participants with prostate cancer. EPIC-26 consists of 26 items under 5 domains. This study will analyze 4 of the domains, including the urinary, bowel, sexual, and hormonal domain. Each domain will be scaled, scored, and compared by arm.
  EPIC-26 assess participant function and bother on a qualitative scale which is then normalized on a scale of 0 to 100 (worst to best) to calculate individual domain scores.
Change in IPSS Score | Baseline, 1 year after treatment
  The "International Prostate Symptom Score" (IPSS) is an eight-question questionnaire that will be administered as a health related quality of life measure for participants with prostate cancer. The IPSS score is reported on a scale of 0 to 35. Scores are broken down as: "Mild" (0 to 7 points), "Moderate" (8 to 19 points), and "Severe" (20 to 35 points). The change in IPSS score from baseline prior to treatment to one year after treatment will be measured.
Change in IPSS Score | Baseline, 3 year after treatment
  The "International Prostate Symptom Score" (IPSS) is an eight-question questionnaire that will be administered as a health related quality of life measure for participants with prostate cancer. The IPSS score is reported on a scale of 0 to 35. Scores are broken down as: "Mild" (0 to 7 points), "Moderate" (8 to 19 points), and "Severe" (20 to 35 points). The change in IPSS score from baseline prior to treatment to three years after treatment will be measured.
Skeletal-related events (SRE) | 5 years after treatment
  Time to the first skeletal-related event is defined as the time from randomization to the first new pathological bone fracture, spinal cord compression, tumor-related orthopedic surgery, and radiation therapy for bone pain. The SRE will be summarized in each arm and compared using Chi-square tests, as well as time-to-event analyses using cumulative incidence methods. The univariable generalized linear models (e.g., Poisson or negative binomial model) will be used to quantify the MDRT effect on the frequency of SRE.

CONTACTS AND LOCATIONS:
Overall Officials: Angela Y Jia, MD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center; Daniel E Spratt, MD, Study Chair — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (2):
- United States (2):
  - University Hospitals Cleveland Medical Center Seidman Cancer Center, Cleveland, Ohio
  - Carbone Cancer Center University of Wisconsin-Madison, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: During study and for 6 months after end of study.
Access Criteria: OnCore, RedCap.